CLINICAL TRIAL: NCT07065422
Title: Comparing Radiomics, Deep Learning, and Fusion Models for Predicting Occult Pleural Dissemination in Patients With Non-small Cell Lung Cancer
Brief Title: AI Models for Predicting Occult Pleural Dissemination in NSCLC
Status: Completed | Type: Observational
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other); Xinqiao hospital of the third military medical university (Unknown)
Responsible Party: Sponsor
Other Study IDs: GUOW
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- non-small cell lung cancer (NSCLC) patients with or without occult pleural dissemination.

SUMMARY:
Occult pleural dissemination (PD) in non-small cell lung cancer (NSCLC) patients is likely to be missed on computed tomography (CT) scans, associated with poor survival, and generally contraindicated for radical surgery. This study aimed to develop and compare the performance of radiomics-based machine learning (ML), deep learning (DL), and fusion models to preoperatively identify occult PDs in NSCLC patients. Patients from three Chinese high-volume medical centers (2016-2023) were retrospectively collected and divided into training, internal test, and external test cohorts. Ten radiomics-based ML models and eight DL models were trained using CT plain scan images at the maximum cross-sectional areas of the primary tumor. Moreover, another two fusion models (prefusion and postfusion) were developed using feature-based and decision-based methods. The receiver operating characteristic curve (ROC) and area under the curve (AUC) were mainly used to compare the predictive performance of the models.

ELIGIBILITY:
Inclusion Criteria:

* pathologically confirmed primary NSCLC with malignant pleural dissemination;
* no preoperative treatment;
* clinicopathological data were complete.

Exclusion Criteria:

* pleural effusion detected preoperatively;
* preoperatively diagnosed with PD;
* poor CT quality or no CT scans within 1 month before surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From January 2016 to December 2023, NSCLC patients with or without surgically confirmed occult PD from three high-volume centers in China were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
The area under the receiver operating characteristic curve (AUC) | through study completion, an average of 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Daping hospital, Chongqing, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code